CLINICAL TRIAL: NCT03952520
Title: Scaling up HIV Prevention Trials Network (HPTN) 074: a Cluster Randomized Implementation Trial of an Evidence-based Intervention for Antiretroviral Therapy for PWID in Vietnam
Brief Title: Scaling up an Evidence-based Intervention for Antiretroviral Therapy for PWID in Vietnam: an Implementation Trial
Acronym: SNaPR01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Ohio State University (Other); Johns Hopkins University (Other); Hanoi Medical University (Other); Vietnam Administration for HIV/AIDS Control (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-2901; 1R01DA047876-01 (NIH); IGHID 11844 (Other: UNC)
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections; Drug Use
Keywords: Cluster randomized controlled implementation trial; Intervention mapping; People who inject drugs; HIV/AIDS; Systems navigation; Psychosocial counseling; Vietnam
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Approach (SA) (Active Comparator): The Standard Approach is a one-size-fits-all multifaceted implementation strategy that was systematically developed using Intervention Mapping.
  Interventions: Other: Standard Approach (SA)
- Tailored Approach (TA) (Experimental): The Tailored Approach includes an implementation strategy that will be tailored to match site-specific barriers to implementation of SNaP at that site.
  Interventions: Other: Tailored Approach (TA)

INTERVENTIONS:
Other: Standard Approach (SA) — The multifaceted implementation strategies for SA sites were identified through centralized Intervention Mapping. Before SNaP implementation starts, the specific set of one-size-fits-all implementation strategies was determined through a formal process with investigators, government stakeholders, and clinical representatives.
  Arms: Standard Approach (SA)
Other: Tailored Approach (TA) — The Tailored Approach includes the multifaceted strategy that will be offered to the Standard Approach condition. It will also be tailored to match site-specific barriers to implementation of SNaP at that site. The strategy for TA sites involves a 2-day site-specific training, monthly coaching calls, and an external technical assistance hotline to help organizations to tailor implementation strategies to address their site-specific needs. At the 2-day TA training, the TA sites will be guided on developing site-specific implementation plans, in which they may use additional implementation strategies that they have identified themselves or selected from a list developed by the central team.
  Arms: Tailored Approach (TA)

SUMMARY:
The purpose of this study is to compare two implementation approaches [Standard Approach (SA) vs. Tailored Approach (TA)] for scaling-up the evidence-based systems navigation and psychosocial counseling integrated intervention (SNaP) in HIV test sites in Vietnam.

DETAILED DESCRIPTION:
This is a cluster randomized, controlled implementation trial to compare two implementation approaches (standard and tailored) for scaling-up the SNaP intervention in 42 HIV test sites in Vietnam. The SNaP intervention combines systems navigation and psychosocial counseling for people who inject drugs (PWID), and it is designed to facilitate PWID's engagement in HIV and substance use care.

The two implementation approaches being compared are:

* Standard Approach (SA); vs.
* Tailored Approach (TA)

SNaP is an evidence-based intervention (EBI) that combines systems navigation and psychosocial counseling to facilitate the engagement of HIV-infected people who inject drugs (PWID) into HIV and substance use care.

The 42 HIV test sites will be randomized in a 1:1 ratio to either the standard approach (SA) procedure or a tailored approach (TA), stratified by engagement of site leadership.

At the HIV test sites, the study will enroll:

* A cohort of 630 PWID who are newly diagnosed or previously diagnosed but not on ART will be enrolled for detailed assessments, including follow-up surveys and dried blood spot collection for viral loads. Additional PWID may be enrolled for medical records assessment without recontact. An additional 242 clinic staff will be enrolled to assess implementation outcomes.
* Note that the original design included ~6200 PWID attending the clinics who consented for medical record assessments only. Upon study initiation, the number of PWID with newly diagnosed HIV infection was substantially lower than predicted. The planned cohort sample was then reduced in size to 630 and all PWID meeting eligibility criteria were referred for enrollment in this cohort.
* HIV test site director boards and staff.

Study activities will span across 5 years, with approximately 27 months at each site and recruitment of PWID participants over 21 months. For the cohort PWID or PWID selected for qualitative interviews, maximum study participation time is 24-27 months. For PWID with medical record assessment only, participation is a one-time visit. For HIV test site director boards and staff, maximum time in the study is 24-27 months.

ELIGIBILITY:
Inclusion Criteria:

PWID participants:

1. HIV infection:

   * Newly diagnosed HIV infection, based on confirmatory test, and not currently on ART at the time of study enrollment; or
   * If previously diagnosed with HIV infection, then must not currently be on ART at the time of study enrollment (self-reported)
2. Age 18 years or older
3. Injection drug use within the past 6 months (self-reported at time of screening)
4. Willing to provide informed consent for the study

Test site director boards and staff:

1. All test site director boards and staff, including the navigators and counselors, at the selected HIV test sites
2. Willing to provide informed consent for the study

Exclusion Criteria:

PWID participants:

1. Residence outside of the catchment area of local antiretroviral therapy (ART) and medication-assisted treatment (MAT, e.g. methadone) clinics
2. Currently on ART at time of study enrollment (self-reported)
3. Planning to move out of the catchment area within the next 24 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian F Go, PhD, MPH, MA, Principal Investigator — University of North Carolina, Chapel Hill; William C Miller, MD, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of an article, after de-identification.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available 6 months to 5 years after publication of the primary outcomes paper.
Access Criteria: Other researchers who provide a methodologically sound proposal to study investigators may be provided access to de-identified data from the study.
  The other researchers must execute a Data Use Sharing Agreement with the University of North Carolina at Chapel Hill (UNC) and obtain the applicable regulatory approvals from their institution before it is permissible for study investigators to share data with the other researchers.

REFERENCES:
- [Derived] Go VF, Giang LM, Phan HTT, Chen JS, Powell BJ, Bartels SM, Nguyen MXB, Sripaipan T, Nong HTT, Dang LTH, Pham MD, Vo SH, Tran HV, Hoang VTH, Nguyen NTK, Chu AV, Levintow SN, Dowdy DW, Sohn H, Pence BW, Miller WC. Scaling an intervention for the engagement of people with HIV who inject drugs into care in Viet Nam: an implementation-effectiveness, cluster-randomised trial. Lancet Glob Health. 2025 Dec;13(12):e2111-e2121. doi: 10.1016/S2214-109X(25)00331-6. PMID 41240949
- [Derived] Nguyen MX, Bartels SM, Akiba CF, Sripaipan T, Nong HT, Dang LT, Tran HV, Hoang VT, Le GM, Go VF, Miller WC, Powell BJ. Tracking modifications to implementation strategies: a case study from SNaP - a hybrid type III randomized controlled trial to scale up integrated systems navigation and psychosocial counseling for PWID with HIV in Vietnam. BMC Med Res Methodol. 2024 Oct 26;24(1):249. doi: 10.1186/s12874-024-02367-3. PMID 39462341
- [Derived] Nguyen MXB, Chu AV, Powell BJ, Tran HV, Nguyen LH, Dao ATM, Pham MD, Vo SH, Bui NH, Dowdy DW, Latkin CA, Lancaster KE, Pence BW, Sripaipan T, Hoffman I, Miller WC, Go VF. Comparing a standard and tailored approach to scaling up an evidence-based intervention for antiretroviral therapy for people who inject drugs in Vietnam: study protocol for a cluster randomized hybrid type III trial. Implement Sci. 2020 Aug 8;15(1):64. doi: 10.1186/s13012-020-01020-z. PMID 32771017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study assessed implementation of the SNaP intervention at 42 HIV Test Sites for 24 months. HIV test site directors and staff were recruited and enrolled prior to SNaP implementation. PWID participants were recruited and enrolled throughout the 24 months of SNaP implementation.
Units Other Than Participants: HIV Test Sites
Groups:
- Standard Approach (SA): The Standard Approach is a one-size-fits-all multifaceted implementation strategy that was systematically developed using Intervention Mapping.
  Standard Approach (SA): The multifaceted implementation strategies for SA sites were identified through centralized Intervention Mapping. Before systems navigation and psychosocial counseling (SNaP) implementation starts, the specific set of one-size-fits-all implementation strategies was determined through a formal process with investigators, government stakeholders, and clinical representatives.
Period: HIV Test Site Directors and Staff
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Started (HIV Test Site Directors and Staff is a distinctly different group than the People Who Inject Drugs (PWID).) | 136; 21 HIV Test Sites | 141; 21 HIV Test Sites
Completed 24-month Survey | 119; 21 HIV Test Sites | 123; 21 HIV Test Sites
Completed | 119; 21 HIV Test Sites | 123; 21 HIV Test Sites
Not Completed | 17; 0 HIV Test Sites | 18; 0 HIV Test Sites
Period: People Who Inject Drugs (PWID)
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Started | 359; 21 HIV Test Sites | 364; 21 HIV Test Sites
Longitudinal Subsample Cohort | 338; 21 HIV Test Sites | 347; 20 HIV Test Sites
Eligible for First Survey | 321; 21 HIV Test Sites | 312; 20 HIV Test Sites
Completed First Survey | 249; 20 HIV Test Sites | 266; 20 HIV Test Sites
Completed | 359; 21 HIV Test Sites | 364; 21 HIV Test Sites
Not Completed | 0; 0 HIV Test Sites | 0; 0 HIV Test Sites

BASELINE CHARACTERISTICS:
Population: Baseline characteristic data were only collected for People Who Inject Drugs (PWID)
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Approach (SA) | Tailored Approach (TA) | Total
Number analyzed (Participants) | 359 | 364 | 723
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [29 to 41] | 37 [32 to 43] | 35 [30 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 31 | 71
  Male | 319 | 333 | 652
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 359 | 364 | 723
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 359 | 364 | 723
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Vietnam | 359 | 364 | 723

OUTCOME MEASURES:

1. Primary Outcome: Fidelity to SNaP Intervention Procedures
Description: Fidelity measures whether the SNaP intervention was delivered as intended.
  Fidelity score = (% Systems navigation sessions completed x Average navigation session quality score) + (% Counseling sessions completed x Average counseling session quality score)
  Session completion will be assessed by reviewing the navigator and counselor logs, while session quality will be assessed by central implementation team review and scoring of a random 10% of all forms (navigation) and audio-recordings (psychosocial counseling). Test site fidelity score range: 0-200 (Higher score indicates higher fidelity.)
Time Frame: Measured over 26 months after SNaP implementation in a clinic
Population: 1 clinic in each arm did not have audio recordings available to calculate the session quality score. Thus, determining a Fidelity score was not possible.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: HIV Test Sites
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Number analyzed (Participants) | 359 | 364
Number analyzed (HIV Test Sites) | 20 | 20
score on a scale | 114.1 (13.5) | 151.4 (21.4)
Statistical Analysis 1: Comparison: Standard Approach (SA) vs Tailored Approach (TA); Test type: Superiority; Mean Difference (Final Values) = 37.3, 95% CI 2-sided [26.5 to 48.1] — This generalized linear model was adjusted for engagement of site leadership. The Standard Approach is the referent

2. Primary Outcome: Percent of PWID Who Initiated ART
Description: Percent of PWID who initiated antiretroviral therapy (ART) among the PWID who initiated SNaP, measured through ART clinic records of consenting PWID and/or self-report.
  This measures ART uptake among PWID who initiated the SNaP intervention.
Time Frame: Medical record reviews conducted within 6 months after enrollment; self-report: 6-12 months after enrollment among those who initiated SNaP
Measure: Number; unit: percentage of participants
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Number analyzed (Participants) | 359 | 364
percentage of participants | 98.6 | 99.5
Statistical Analysis 1: Comparison: Standard Approach (SA) vs Tailored Approach (TA); Test type: Superiority; Risk Difference (RD) = 2.0, 95% CI 2-sided [2.0 to 2.1] — This generalized linear model was adjusted for engagement of site leadership and used generalized estimating equations to account for clustering by HIV test site. The Standard Approach is the referent

3. Secondary Outcome: Percent of PWID Who Were Contacted and Participated in SNaP
Description: Penetration of SNaP at the test sites is assessed by this measure. Penetration of SNaP is defined as the proportion of newly diagnosed or previously diagnosed and not currently on ART PWID at test sites who are contacted by a navigator and/or counselor and participate in a SNaP session.
  Penetration of SNaP will be assessed at 12 and 24 months after implementation of SNaP in a clinic. Only the 24-month assessment is reported.
Time Frame: Up to 24 months after implementation of SNaP in a clinic
Measure: Number; unit: percentage of participants
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Number analyzed (Participants) | 359 | 364
percentage of participants | 100 | 100

4. Secondary Outcome: Mean Acceptability Score of SNaP by PWID (AIM)
Description: Acceptability is the perception that the SNaP intervention is agreeable, palatable, or satisfactory to PWID. Acceptability among PWID participants will be assessed using the Acceptability of Intervention Measure (AIM), which consists of 4 items containing responses on a 5-point Likert scale. The AIM score will be the sum of the 4 item responses ranging from 4-20. Higher AIM scores indicate higher acceptability. Acceptability of SNaP by PWID will be assessed at 12, 18, and 24 months after SNaP implementation in a clinic. Only the first acceptability assessment collected for a participant is reported.
Time Frame: Up to 24 months after SNap implementation in a clinic
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Number analyzed (Participants) | 249 | 266
score on a scale | 16.7 (1.1) | 16.8 (1.3)
Statistical Analysis 1: Comparison: Standard Approach (SA) vs Tailored Approach (TA); Test type: Superiority; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.4] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Mean Acceptability Score of SNaP by Test Site Staff (OADRI)
Description: Acceptability is the perception that the SNaP intervention is agreeable, palatable, or satisfactory to test site staff. Acceptability among site staff will be assessed using the Ottawa Acceptability of Decision Rules Instrument (OADRI), a 12-item scale, staff and client acceptability of an innovation in a clinic setting. Eight of the 12 items were included in the assessment, excluding 4 irrelevant questions for the study setting. Scores range from 8-48. Higher OADRI scores indicate higher acceptability. Acceptability of SNaP by Test Site Staff will be assessed at 12 and 24 months after SNaP implementation in a clinic. Only the 24-month assessment is reported.
Time Frame: 24 months after implementation of SNaP in a clinic
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Number analyzed (Participants) | 119 | 123
score on a scale | 37.7 (5.1) | 37.1 (7.0)
Statistical Analysis 1: Comparison: Standard Approach (SA) vs Tailored Approach (TA); Test type: Superiority; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-3.1 to 2.0] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Percent of PWID Who Are Virally Suppressed
Description: Percent of PWID who are virally suppressed among the PWID who initiated SNaP. Viral suppression is defined as <1000 copies/mL. (This outcome will be measured only in the PWID subsample cohort.) Percent of PWID virally suppressed will be assessed at 12, 18, and 24 months after SNaP implementation in a clinic. Only the first assessment collected for a participant is reported.
Time Frame: Up to 24 months after implementation of SNaP in a clinic
Measure: Number; unit: percentage of participants
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Number analyzed (Participants) | 321 | 312
percentage of participants | 43.0 | 59.3
Statistical Analysis 1: Comparison: Standard Approach (SA) vs Tailored Approach (TA); Test type: Superiority; Prevalence Difference = 15.8, 95% CI 2-sided [5.0 to 26.5] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Percent of PWID on Medication-Assisted Treatment (MAT)
Description: Percent of PWID alive and on MAT among the PWID who initiated SNaP, measured through medical records and/or self-report of consenting PWID. This measures MAT uptake among PWID who initiated SNaP. Percent of PWID on MAT will be assessed at 12, 18, and 24 months after SNaP implementation in a clinic. Only the first assessment collected for a participant is reported.
Time Frame: Up to 24 months after SNaP implementation in a clinic
Measure: Number; unit: percentage of participants
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Number analyzed (Participants) | 321 | 312
percentage of participants | 10.9 | 12.8
Statistical Analysis 1: Comparison: Standard Approach (SA) vs Tailored Approach (TA); Test type: Superiority; Prevalence Difference = 1.6, 95% CI 2-sided [-6.9 to 10.0] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Incremental Cost-Effectiveness Ratio of SA Compared to TA for SNaP Implementation
Description: The incremental cost per incremental ART uptake, comparing TA to SA, measured as: The difference in costs of implementing SNaP in TA compared to SA sites divided by the difference in ART uptake in TA compared to SA sites.
  Incremental cost-effectiveness of SNaP implementation will be assessed up to 24 months after SNaP implementation in a clinic.
Time Frame: Up to 24 months after SNaP implementation in a clinic.
Measure: Number; unit: USD/Incremental Person Initiating ART
Groups:
- Tailored Approach (TA) vs Standard Approach (SA): The Tailored Approach includes an implementation strategy that will be tailored to match site-specific barriers to implementation of SNaP at that site.
  Tailored Approach (TA): The Tailored Approach includes the multifaceted strategy that will be offered to the Standard Approach condition. It will also be tailored to match site-specific barriers to implementation of SNaP at that site. The strategy for TA sites involves a 2-day site-specific training, monthly coaching calls, and an external technical assistance hotline to help organizations to tailor implementation strategies to address their site-specific needs. At the 2-day TA training, the TA sites will be guided on developing site-specific implementation plans, in which they may use additional implementation strategies that they have identified themselves or selected from a list developed by the central team.
  The Standard Approach is a one-size-fits-all multifaceted implementation strategy that was systematically developed using Intervention Mapping.
  Standard Approach (SA): The multifaceted implementation strategies for SA sites were identified through centralized Intervention Mapping. Before SNaP implementation starts, the specific set of one-size-fits-all implementation strategies was determined through a formal process with investigators, government stakeholders, and clinical representatives.
Arm/Group | Tailored Approach (TA) vs Standard Approach (SA)
Number analyzed (Participants) | 723
USD/Incremental Person Initiating ART | 25,872.75

9. Secondary Outcome: Percent of PWID Alive and Remaining on ART
Description: Percent of PWID alive and on ART among the PWID who initiated SNaP, measured through medical records and/or self-report of consenting PWID. Percent of PWID alive and remaining on ART will be assessed at 12, 18, and 24 months after SNaP implementation in a clinic. Only the first assessment collected for a participant is reported.
Time Frame: Up to 24 months after SNaP implementation in a clinic
Measure: Number; unit: percentage of participants
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Number analyzed (Participants) | 321 | 312
percentage of participants | 74.5 | 84.3
Statistical Analysis 1: Comparison: Standard Approach (SA) vs Tailored Approach (TA); Test type: Superiority; Prevalence Difference = 6.2, 95% CI 2-sided [-1.5 to 13.8] — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Percent of Clinics Continuing to Offer SNaP After Completion of Study Activities
Description: Sustainment of SNaP at the test sites is assessed by this measure.
  Sustainment of SNaP is defined as the % of clinics continuing to offer SNaP after completion of study activities, based on survey of clinic staff
  Sustainment of SNaP will be assessed up to 37 months after SNaP implementation in a clinic.
Time Frame: Up to 37 months after SNaP implementation in a clinic
Population: HIV Test Site Directors and Staff who completed a sustainment survey 6-10 months following the completion of the SNaP activities at each site.
Measure: Number; unit: % of Clinics
Units Other Than Participants: Clinics
Arm/Group | Standard Approach (SA) | Tailored Approach (TA)
Number analyzed (Participants) | 111 | 107
Number analyzed (Clinics) | 21 | 21
% of Clinics | 33 | 57

ADVERSE EVENTS:
Time Frame: Adverse events were collected for HIV Test Site Directors and Staff and the longitudinal subsample cohort of PWID from the time of signing informed consent until the respective site at which the participant was enrolled reached implementation Month 24, up to approximately 24 months. Adverse events were collected for PWID participants not in the longitudinal subsample cohort from the time of signing informed consent until the completion of intervention activities, up to approximately 8 weeks.
Groups:
- Standard Approach (SA) PWID: PWID enrolled at clinics implementing SNaP under the Standard Approach.
- Tailored Approach (TA) PWID: PWID enrolled at clinics implementing SNaP under the Tailored Approach.
- Standard Approach (SA) HIV Test Site Directors and Staff: HIV Test Site Directors and Staff working at clinics implementing SNaP under the Standard Approach.
- Tailored Approach (TA) HIV Test Site Directors and Staff: HIV Test Site Directors and Staff working at clinics implementing SNaP under the Tailored Approach.
Arm/Group | Standard Approach (SA) PWID | Tailored Approach (TA) PWID | Standard Approach (SA) HIV Test Site Directors and Staff | Tailored Approach (TA) HIV Test Site Directors and Staff
All-Cause Mortality (participants affected / at risk) | 23/359 | 42/364 | 0/136 | 0/141
Serious Adverse Events (participants affected / at risk) | 0/359 | 0/364 | 0/136 | 0/141
Other Adverse Events (participants affected / at risk) | 0/359 | 0/364 | 0/136 | 0/141

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT03952520/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT03952520/ICF_000.pdf